CLINICAL TRIAL: NCT05718128
Title: Clinical Study of Endocardial Myocardial Biopsy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0131
Record Dates: First submitted 2021-06-15; First posted 2023-02-08 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-01

CONDITIONS: Myocarditis; Cardiomyopathies; Heart Failure; Cardiac Tumor; Endocardiomyocardial Biopsy
MeSH Terms: conditions — Myocarditis; Cardiomyopathies; Heart Failure; Heart Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biopsy (Experimental): patients
  Interventions: Procedure: Endocardiomyocardial biopsy

INTERVENTIONS:
Procedure: Endocardiomyocardial biopsy — Endocardiomyocardial biopsy

SUMMARY:
In this study, patients with endocardial myocardial biopsy were selected to observe the safety of the operation, and pathological examination was performed. If necessary, special tests such as viral examination, mass spectrometry and molecular biology were performed to confirm the diagnosis, and follow-up was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no gender restriction, age 18-80 years old, receiving endocardial myocardial biopsy in the Second Affiliated Hospital of Zhejiang University School of Medicine;
* Patients with myocarditis, cardiomyopathy, heart failure and cardiac tumor of unknown clinical cause;
* Have the ability to understand the test, can cooperate with investigators.

Exclusion Criteria:

* Unable to understand or unwilling to fill in informed consent forms or follow visitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE-4 | 10 year
  incidences of MACE-4(cardiovascular death, myocardial infarction, stroke and hospitalized unstable angina)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China